CLINICAL TRIAL: NCT01935934
Title: A Phase 2 Study of XL184 (Cabozantinib) in Recurrent or Metastatic Endometrial Cancer
Brief Title: Cabozantinib S-Malate in Treating Patients With Recurrent or Metastatic Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00890; NCI-2013-00890 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHL-086; 9322 (Other: University Health Network-Princess Margaret Hospital); 9322 (Other: CTEP); N01CM00032 (NIH); N01CM00038 (NIH); N01CM00071 (NIH); UM1CA186644 (NIH); NCT01815151 (obsolete NCT alias)
Record Dates: First submitted 2013-09-03; First posted 2013-09-05 (Estimated); Results first posted 2020-07-14 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Endometrial Adenosquamous Carcinoma; Endometrial Clear Cell Adenocarcinoma; Endometrial Mixed Cell Adenocarcinoma; Endometrial Serous Adenocarcinoma; Metastatic Endometrioid Adenocarcinoma; Recurrent Malignant Uterine Corpus Neoplasm; Stage IV Uterine Corpus Carcinoma or Carcinosarcoma by AJCC v7 Stage; Stage IVA Uterine Corpus Carcinoma or Carcinosarcoma by AJCC v7 Stage; Stage IVB Uterine Corpus Carcinoma or Carcinosarcoma by AJCC v7 Stage; Uterine Corpus Carcinosarcoma
MeSH Terms: conditions — Carcinoma, Endometrioid | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (cabozantinib s-malate) (Experimental): Patients receive 60 mg cabozantinib s-malate PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib S-malate; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL 184; XL-184; XL184
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well cabozantinib s-malate works in treating patients with endometrial cancer that has come back (recurrent) or has spread to other places in the body (metastatic). Cabozantinib s-malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine efficacy of single agent cabozantinib s-malate (cabozantinib) in women previously receiving one line of chemotherapy for metastatic endometrial cancer or with progression within 12 months of completing adjuvant therapy, with co-primary endpoints of objective response rate by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and progression-free-survival at 12 weeks (PFS).

SECONDARY OBJECTIVES:

I. Correlation of clinical response with baseline molecular status of archival tumor (hepatocyte growth factor receptor [c-met] amplification & mutation status) and overall survival.

OUTLINE:

Patients receive cabozantinib s-malate orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 4 weeks or every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic endometrial cancer; eligible histologies for the experimental cohort are: endometrioid or serous; eligible histologies for the exploratory cohort are: carcinosarcoma, clear cell, mixed, adenosquamous and any other rare sub-type of endometrial cancer
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 10 mm with computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam and >= 15 mm in short axis for nodal lesions; patients must have radiographic evidence of disease progression following the most recent line of treatment
* Prior therapy: Eligible subjects must have had 1 line of systemic cytotoxic treatment; this may be adjuvant therapy with documented progression within 12 months of completion, or 1 line of cytotoxic therapy for metastatic disease; NOTE: eligible patients are allowed up to 2 lines of systemic cytotoxic treatment, of which only 1 line is allowed for metastatic disease; the acceptance of progression within 12 months of adjuvant is part inclusion to not require patient to re-challenge with chemotherapy (chemo) if they progressed soon after adjuvant therapy; prior hormonal therapy for metastatic/recurrent disease is also allowed; prior targeted therapy not directed against cMET or vascular endothelial growth factor (VEGF) pathways is allowed
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 3 months
* Absolute neutrophil count >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 X institutional upper limit of normal
* Creatinine =< 1.5 x ULN OR creatinine clearance >= 50 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Hemoglobin >= 90 g/L
* Serum albumin >= 28 g/L
* Lipase < 2.0 x ULN; no radiologic/clinical evidence of pancreatitis
* Urine protein/creatinine ratio (UPCR) =< 1
* Serum phosphorus, calcium, magnesium and potassium >= lower limit of normal (LLN)
* Women of childbearing potential must have a negative pregnancy test at screening; women of childbearing potential include women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are not postmenopausal; postmenopausal is defined as amenorrhea >= 12 consecutive months; note: women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, ovarian suppression or any other reversible reason
* Women of child-bearing potential must agree to use adequate contraception prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately; sexually active subjects must agree to use medically accepted barrier methods of contraception (e.g., male or female condom) during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used; all subjects of reproductive potential must agree to use both a barrier method and a second method of birth control during the course of the study and for 4 months after the last dose of study drug(s)
* Patients must consent to analysis on archival tissue; if archival sample is not available, a sufficient tumor biopsy can be performed a minimum of 28 days prior to start of treatment if felt to be clinically reasonable
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy (including investigational cytotoxic chemotherapy), biologic agents (e.g., cytokines or antibodies) or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) before the first dose of study treatment or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Prior treatment with cabozantinib
* The subject has received radiation therapy:

  * To bone metastasis within 14 days before the first dose of study treatment
  * To any other site(s) within 28 days before the first dose of study treatment
* The subject has received radionuclide treatment within 6 weeks of the first dose of study treatment
* The subject has received prior treatment with a small molecule kinase inhibitor or a hormonal therapy (including investigational kinase inhibitors or hormones) within 14 days or five half-lives of the compound or active metabolites, whichever is longer, before the first dose of study treatment
* The subject has received any other type of investigational agent within 28 days before the first dose of study treatment
* The subject has not recovered to baseline or Common Terminology Criteria for Adverse Events (CTCAE) =< grade 1 from related toxicity to all prior therapies except alopecia and other non-clinically significant adverse events (AEs)
* Any other prior malignancy from which the patient has been disease free for less than 3 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of any site or any other cancer
* Patients with known brain metastases should be excluded from this clinical trial
* The subject has prothrombin time (PT)/international normalized ratio (INR) or partial thromboplastin time (PTT) test >= 1.3 x the laboratory ULN =< 7 days before the first dose of study treatment
* Therapeutic anticoagulation with warfarin, antiplatelet agents (e.g., clopidogrel), thrombin, or Factor Xa inhibitors is not allowed; therapeutic anticoagulation with low molecular weight heparin (LMWH) is allowed as well as prophylactic anticoagulation using low dose aspirin (=< 81 mg/day), low-dose warfarin (=< 1 mg/day), and LMWH
* The subject requires chronic concomitant treatment of strong CYP3A4 inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital, and St. John's wort)
* The subject has experienced any of the following:

  * Clinically-significant gastrointestinal bleeding within 6 months before the first dose of study treatment
  * Hemoptysis of >= 0.5 teaspoon (2.5 mL) of red blood within 3 months before the first dose of study treatment
  * Any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment
* The subject has tumor in contact with, invading or encasing any major blood vessels
* The subject has evidence of tumor invading the gastrointestinal (GI) tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders including:

    * Congestive heart failure (CHF): New York Heart Association (NYHA) class III (moderate) or class IV (severe) at the time of screening
    * Concurrent uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mmHg systolic, or > 90 mmHg diastolic despite optimal antihypertensive treatment within 7 days of the first dose of study treatment
    * Any history of congenital long QT syndrome
    * Any of the following within 6 months before the first dose of study treatment:

      * Unstable angina pectoris
      * Clinically-significant cardiac arrhythmias
      * Stroke (including transient ischemic attack [TIA], or other ischemic event)
      * Myocardial infarction
      * Thromboembolic event requiring therapeutic anticoagulation (note: subjects with a venous filter [e.g. vena cava filter] are not eligible for this study)
* Gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation including:

  * Any of the following within 28 days before the first dose of study treatment

    * Intra-abdominal tumor/metastases invading GI mucosa
    * Active peptic ulcer disease,
    * Inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis
    * Malabsorption syndrome
  * Any of the following within 6 months before the first dose of study treatment:

    * Abdominal fistula
    * Gastrointestinal perforation
    * Bowel obstruction or gastric outlet obstruction
    * Intra-abdominal abscess; note: complete resolution of an intra-abdominal abscess must be confirmed prior to initiating treatment with cabozantinib even if the abscess occurred more than 6 months before the first dose of study treatment
* Other disorders associated with a high risk of fistula formation including percutaneous endoscopic gastrostomy (PEG) tube placement within 3 months before the first dose of study therapy
* Other clinically significant disorders such as:

  * Active uncontrolled infection requiring intravenous systemic treatment within 14 days before the first dose of study treatment
  * Serious non-healing wound/ulcer/bone fracture within 28 days before the first dose of study treatment
  * History of organ transplant
  * Concurrent uncompensated hypothyroidism or thyroid dysfunction within 7 days before the first dose of study treatment
  * History of major surgery as follows:

    * Major surgery within 3 months of the first dose of cabozantinib if there were no wound healing complications or within 6 months of the first dose of cabozantinib if there were wound complications
    * Minor surgery within 1 month of the first dose of cabozantinib if there were no wound healing complications or within 3 months of the first dose of cabozantinib if there were wound complications

      * In addition, complete wound healing from prior surgery must be confirmed at least 28 days before the first dose of cabozantinib irrespective of the time from surgery
* The subject is unable to swallow tablets
* The subject has a corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms =< 7 days before the first dose of study treatment
* The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to XL184
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with XL184
* Known human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2013-05-08 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2024-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neesha Dhani, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (19):
- United States (12):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - City of Hope South Pasadena, South Pasadena, California
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
- Canada (7):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Dhani NC, Hirte HW, Wang L, Burnier JV, Jain A, Butler MO, Welch S, Fleming GF, Hurteau J, Matsuo K, Matei D, Jimenez W, Johnston C, Cristea M, Tonkin K, Ghatage P, Lheureux S, Mehta A, Quintos J, Tan Q, Kamel-Reid S, Ludkovski O, Tsao MS, Wright JJ, Oza AM. Phase II Trial of Cabozantinib in Recurrent/Metastatic Endometrial Cancer: A Study of the Princess Margaret, Chicago, and California Consortia (NCI9322/PHL86). Clin Cancer Res. 2020 Jun 1;26(11):2477-2486. doi: 10.1158/1078-0432.CCR-19-2576. Epub 2020 Jan 28. PMID 31992589

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental (Endometriod + Serous); Exploratory (Uncommon Histology): Patients receive cabozantinib s-malate PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
Period: Overall Study
Arm/Group | Experimental (Endometriod + Serous) | Exploratory (Uncommon Histology)
Started | 70 | 32
Completed | 70 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental (Endometriod + Serous) | Exploratory (Uncommon Histology) | Total
Number analyzed (Participants) | 70 | 32 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 14 | 47
  >=65 years | 37 | 18 | 55
Age, Continuous [Median (Full Range); unit: years] | 70 [38 to 84] | 66 [25 to 75] | 66 [25 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 32 | 102
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 67 | 27 | 94
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 9 | 4 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 54 | 25 | 79
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 48 | 22 | 70
  United States | 22 | 10 | 32

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: At 12 weeks, then every 8 weeks during treatment; up to 12 weeks post-treatment if discontinued due to toxicities, a maximum of 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental (Endometriod + Serous) | Exploratory (Uncommon Histology)
Number analyzed (Participants) | 70 | 32
Participants | 9 | 2

2. Primary Outcome: Progression-free Survival
Description: Defined as the percentage of patients progression free 12 weeks from starting treatment.
Time Frame: Time from start of treatment to time of progression or death, assessed at 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Experimental (Endometriod + Serous) | Exploratory (Uncommon Histology)
Number analyzed (Participants) | 70 | 32
percentage of participants | 67.17 | 46.88
Statistical Analysis 1: Comparison: Experimental (Endometriod + Serous); Test type: Other; Trial design discriminated between co-primary endpoints of objective RR of 30% (vs 10%) and 12-week PFS of 55% (vs 30%). The design had 86% power to detect a true objective RR of at least 30% and at least 90% power to detect a true 12-week PFS rate of atleast 55% (or a median PFS of 3.4 months). The parallel exploratory cohort of uncommon histology cancers was analyzed independently

3. Secondary Outcome: Number of Participants With Archival Specimens That Had C-met Amplification or Mutation
Description: Will correlate with clinical response.
  83 tumors were profiled on the NGS TruSeq amplicon panel and 1 on Sequenom. Fields with at least 50 tumor cells were captured to analyze 100 non-overlapping tumor cell nuclei to calculate a ratio of MET to CEP7 signal; MET ampliction was defined as MET/CEP7 ratio >=2.
Time Frame: Baseline
Population: Archival tumor was available in 91 patients. Genomic analysis failed in 7. Of the remaining 84, 83 tumors were profiled on the NGS TruSeq amplicon panel and 1 on Sequenom to analyze the number of mutations observed.
Measure: Number; unit: participants
Groups:
- Endometrioid; Serous; Carcinosarcoma; Other Histology: Patients receive 60 mg cabozantinib s-malate PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
Arm/Group | Endometrioid | Serous | Carcinosarcoma | Other Histology
Number analyzed (Participants) | 31 | 30 | 15 | 8
participants
  PTEN | 13 | NA — Below level of detection | NA — Below level of detection | NA — Below level of detection
  PIK3CA | 10 | 10 | 6 | NA — Below level of detection
  CTNNB1 | 9 | NA — Below level of detection | NA — Below level of detection | NA — Below level of detection
  KRAS | 8 | 3 | 3 | NA — Below level of detection
  TP53 | 6 | 19 | 7 | NA — Below level of detection
  MET | 0 | 0 | 0 | NA — Below level of detection

4. Secondary Outcome: Overall Survival
Description: Will correlate with clinical response.
Time Frame: Time from start of treatment to time of death, every 6 months
Population: Participants followed for overall survival, every 6 months until death
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental (Endometriod + Serous) | Exploratory (Uncommon Histology)
Number analyzed (Participants) | 6 | 7
Participants | 4 | 3

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 6 months with a maximum of up to 4 years.
Description: As pre-defined in the study protocol, adverse events were collected and analyzed for both cohorts together (combined data).
Groups:
- Treatment (Cabozantinib S-malate): Patients receive cabozantinib s-malate PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
Arm/Group | Treatment (Cabozantinib S-malate)
All-Cause Mortality (participants affected / at risk) | 7/102
Serious Adverse Events (participants affected / at risk) | 42/102
Other Adverse Events (participants affected / at risk) | 102/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cabozantinib S-malate) (N=102)
Gastric hemorrhage (Gastrointestinal disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 4 (5)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Death (General disorders) | 2 (2)
Gastrointestinal fistula (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Akathisia (Nervous system disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (5)
Fever (General disorders) | 2 (2)
Colonic perforation (Gastrointestinal disorders) | 4 (4)
Alanine aminotransferase increased (Investigations) | 3 (3)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Vascular disorders) | 6 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Colonic fistula (Gastrointestinal disorders) | 2 (2)
Dental caries (Gastrointestinal disorders) | 1 (1)
Ileal perforation (Gastrointestinal disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lipase increased (Investigations) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Blood (Infections and infestations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
GGT increased (Investigations) | 1 (2)
Abdominal infection (Infections and infestations) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cabozantinib S-malate) (N=102)
Fatigue (General disorders) | 65 (65)
Anorexia (Metabolism and nutrition disorders) | 49 (49)
Weight loss (Investigations) | 31 (31)
Hypertension (Vascular disorders) | 52 (52)
Diarrhea (Gastrointestinal disorders) | 60 (60)
Nausea (Gastrointestinal disorders) | 46 (46)
Dysgeusia (Gastrointestinal disorders) | 42 (42)
Mucositis (Gastrointestinal disorders) | 38 (38)
Vomiting (Gastrointestinal disorders) | 19 (19)
Gastrointestinal reflux (Gastrointestinal disorders) | 17 (17)
Dyspepsia (Gastrointestinal disorders) | 13 (13)
Dry mouth (Gastrointestinal disorders) | 15 (15)
Abdominal pain (Gastrointestinal disorders) | 19 (19)
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 40 (40)
Dry skin (Skin and subcutaneous tissue disorders) | 11 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (12)
Anemia (Blood and lymphatic system disorders) | 27 (27)
White blood cell decreased (Investigations) | 33 (33)
Lymphocyte count decreased (Investigations) | 31 (31)
Neutrophil count decreased (Investigations) | 23 (23)
Platelet count decreased (Investigations) | 20 (20)
Aspartate aminotransferase increased (Investigations) | 66 (66)
Hypomagnesemia (Investigations) | 48 (48)
Hypophosphatemia (Investigations) | 30 (30)
Alkaline aminotransferase increased (Investigations) | 24 (24)
Hypoalbuminemia (Investigations) | 29 (29)
GGT increased (Investigations) | 17 (17)
Hyponatremia (Investigations) | 21 (21)
Hypokalemia (Investigations) | 19 (19)
Blood bilirubin increased (Investigations) | 12 (12)
Proteinuria (Renal and urinary disorders) | 12 (12)
Endocrine disorder (Endocrine disorders) | 12 (12) — Hypo/Hyperthyroidism
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 15 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (11)
Headache (Nervous system disorders) | 11 (11)
Vascular disorder (Vascular disorders) | 12 (12) — Bleeding
Venous thromboembolism (Vascular disorders) | 11 (11)
Gastrointestinal disorder (Gastrointestinal disorders) | 8 (8) — GI perforation/fistula
Alanine aminotransferase increased (Investigations) | 64 (64)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT01935934/Prot_SAP_000.pdf